CLINICAL TRIAL: NCT03114839
Title: The Effect of Daily Consumption of a Probiotic Drink Containing Lactobacillus Casei Strain Shirota on the Small Intestinal Microbiota in Healthy Male Subjects as Measured by the IntelliCap Sampling Capsule System.
Brief Title: Effect of Lactobacillus Casei Shirota on the Small Intestinal Microbiota (ROBIN)
Acronym: ROBIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yakult Honsha European Research Center, ESV (Other)
Collaborators: NIZO Food Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL59320.081.16
Record Dates: First submitted 2017-04-10; First posted 2017-04-14 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: Lactobacillus casei strain Shirota; Yakult; IntelliCap

STUDY DESIGN:
Intervention Model Description: The study is a dietary intervention study with a repeated measures design, comparing the upper gastrointestinal microbiota profiles in healthy male subjects before and after consumption of a probiotic drink containing Lactobacillus casei strain Shirota.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary Supplement: Lactobacillus casei strain Shirota (LcS) (Experimental)
  Interventions: Dietary Supplement: Lactobacillus casei strain Shirota (LcS)

INTERVENTIONS:
Dietary Supplement: Lactobacillus casei strain Shirota (LcS) — A fermented milk containing LcS, 65 ml for oral administration, 1 bottle per day for 7 days. One bottle of the drink contains: 42.9 kcal/182 kJ; less than 0.1 g of fat; 9.6 g of carbohydrate; 0.01 g of sodium; 0.9 g of protein; and at least 6.5 x 10^9 colony-forming units of LcS.
  Other Names: Commercial name: Yakult®

SUMMARY:
Currently, obtaining samples directly from the small bowel is difficult due to the highly invasive intubation methods used. Research on the effect of dietary probiotics on the gut microbiota is therefore largely dependent on measurement of the microbial composition in fecal samples. At best, the measurement in fecal samples reflects microbial composition of the large intestine. The microbial composition in the small intestine differs substantially from the composition in feces. In addition, many physiological processes that are modulated by dietary probiotics, such as immunoregulation, mainly occur in the small intestine. Therefore, it is vital to study the effects of dietary probiotics on the small intestinal microbiota, as well. Successful sampling of the small intestine has been demonstrated in animals and humans, using the IntelliCap® CR system. The main aim of the current study is to explore and compare the small intestinal microbiota profiles in healthy subjects before and after consumption of a probiotic drink containing Lactobacillus casei strain Shirota (LcS) (Yakult®).

DETAILED DESCRIPTION:
The study is a dietary intervention study with a repeated measures design, comparing the upper gastrointestinal microbiota profiles in healthy male subjects before and after consumption of a probiotic drink containing LcS.

This study is explorative in nature. This pilot-study is used to explore trends in microbiota profile shifts in the small intestine. In addition, the investigators would like to explore whether these microbial shifts are similar to those observed in fecal samples. Information derived from this pilot-study can be used to design future intervention studies focusing on either the effect of probiotics on microbial shifts in the small or large intestine.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Age 18-30yrs
3. BMI between 18,5-25 kg/m2
4. Healthy as assessed by the NIZO lifestyle and health questionnaire ("Verklaring leefgewoonten en gezondheid").
5. Non-smoking
6. Regular bowel movement (defecation on average once a day, at least 4 times/week).
7. Signed informed consent
8. Access to internet
9. Access to freezer for storage of biological samples
10. Voluntary participation
11. Willing to accept disclosure of the financial benefit of participation in the study to the authorities concerned.
12. Willing to accept use of all encoded data, including publication, and the confidential use and storage of all data for the study for at least 15 years.
13. Willing to accept information-transfer concerning participation in the study, or information regarding health, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from his general practitioner.
14. Willing to comply with study procedures.

Exclusion Criteria:

1. Alcohol consumption > 15 units/week and > 3/day.
2. Allergic to dairy products (milk allergy or lactose intolerance).
3. Carrying a pacemaker or any other (implanted) medical electronic device.
4. Drug abuse.
5. Having diarrhea within two (2) months prior to the study start.
6. Heavy exercise or sports training > 10 hours/week.
7. History or presence of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
8. Mental status that is incompatible with the proper conduct of the study.
9. Participation in any scientific study with oral, intravenous or inhalatory administration of any substances during two (2) months before study start.
10. Presence of swallowing disorder or problems with gastro-intestinal transit.
11. Reported special diets such as vegetarian, vegan, or macrobiotic.
12. Scheduled for an MRI scan during the study period.
13. Unstable body weight (weight gain or loss >5kg in the past three (3) months).
14. Use of antibiotics during the six (6) months prior to study start.
15. Use of any prescribed or non-prescribed medication (other than paracetamol) during the three (3) weeks prior to study start.
16. Use of laxatives and probiotic, prebiotic and fiber supplements during the two (2) months prior to study start.
17. Personnel of research institute(s) involved in execution of the study, their partner and their first and second degree relatives
18. Not having a general practitioner
19. Not willing to have an X-ray if the capsule is not recovered from the feces.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2017-09-04 (Estimated); Primary Completion 2017-10-31 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
Microbiota composition in the small intestine | 7 days after consuming a probiotic drink containing Lactobacillus casei strain Shirota (LcS)
  Relative abundance of microbiota species (% of total) in the small intestine

SECONDARY OUTCOMES:
Microbiota composition in feces | 7 days after consuming a probiotic drink containing LcS
  Relative abundance of microbiota species (% of total ) in feces
LcS recovery | 7 days after consuming a probiotic drink containing LcS
  LcS recovery in the small intestine and feces
Stool habits | 7 days after consuming a probiotic drink containing LcS
  Effect of LcS on stool frequency, stool consistency and gastrointestinal symptoms

OTHER OUTCOMES:
Biomarkers | 7 days after consuming a probiotic drink containing LcS
  Feasibility assessment of measuring potential biomarkers in the small intestine and feces

CONTACTS AND LOCATIONS:
Locations (1):
- NIZO Food Research, Ede, Utrecht,, Netherlands

IPD SHARING:
Plan to Share IPD: No